CLINICAL TRIAL: NCT00989807
Title: Expanded Access for Aztreonam Lysine for Inhalation in Canadian Patients With Cystic Fibrosis and Pseudomonas Aeruginosa Airway Infection Who Have Limited Treatment Options and Are at Risk for Disease Progression
Brief Title: Expanded Access Program for Aztreonam Lysine for Inhalation in Canadian Patients With Cystic Fibrosis
Acronym: EAP
Status: Approved for marketing | Type: Expanded Access
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: EA-US-205-0122
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-10

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa
Keywords: CF; Cystic fibrosis; Pseudomonas aeruginosa; EAP; Expanded access; AZLI; Aztreonam lysine
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

INTERVENTIONS:
Drug: Aztreonam lysine — Open-label, expanded access for Aztreonam lysine for inhalation 75 mg three times daily

SUMMARY:
This program is to provide expanded access to aztreonam lysine for inhalation (AZLI) prior to its commercial availability to patients with cystic fibrosis (CF) and chronic P. aeruginosa airway infection who have limited treatment options and are at risk for disease progression.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 years of age
* Patient has CF as diagnosed by one of the following:
* Documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test, or
* Two well characterized genetic mutations in the CFTR gene, or
* Abnormal nasal potential difference with accompanying symptoms characteristic of CF
* PA present in expectorated sputum or throat swab culture within 2 months prior to consent
* Patient must be able to provide written informed consent/assent prior to any study related procedure; parent/guardian must be able to give written informed consent as necessary prior to any study related procedure
* At high risk for disease progression as defined by one of the following patient populations:
* FEV1 ≤ 50 % predicted at the time of consent OR
* Completed participation in CP-AI-006 (through Visit 20). Patients who withdraw from CP-AI-006 prior to completing all courses of AZLI and all study visits will not be eligible for this protocol.

Exclusion Criteria:

* Patients with any serious or active medical or psychiatric illness that, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol or dosing requirements
* Patients with hypersensitivity to any of the components of the drug product
* Currently enrolled in another clinical trial
* Pregnant or lactating females

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - University of Calgary, Adult CF Clinic, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Michael's Hospital, Toronto, Ontario
  - Centre de Recherche du CHUM, Montreal, Quebec